CLINICAL TRIAL: NCT04709172
Title: Prospective, Non-controlled Pilot Study to Evaluate the Efficacy and Safety of Cefditoren Pivoxil in COVID-19 Patients With Mild to Moderate Pneumonia
Brief Title: Pilot Study of Cefditoren Pivoxil in COVID-19 Patients With Mild to Moderate Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meiji Pharma Spain S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPS-ME1207/401
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-01

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; pneumonia; cefditoren; outpatient
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — cefditoren pivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cefditoren pivoxil 400mg (Experimental): Cefditoren pivoxil 400mg bid for 7 days
  Interventions: Drug: Cefditoren pivoxil 400mg

INTERVENTIONS:
Drug: Cefditoren pivoxil 400mg — Cefditoren pivoxil 400mg bid for 7 days
  Other Names: CDN-PI 400mg

SUMMARY:
The global pandemic of novel coronavirus disease 2019 (COVID-19) began in Wuhan, China, in December 2019, and has since spread worldwide. The disease is mild in 85% of cases but the remaining 15% requires hospitalization and/or intensive care.

Recent publications show that a significant number of COVID-19 patients are co-infected with one or more pathogens. Most co-infections occurred within 1-4 days of onset of COVID-19 disease and a considerable number of patients arrive to the Emergency rooms with mild-moderate respiratory symptoms compatible with pneumonia of presumed bacterial origin and not severe enough for requiring hospitalization. It therefore seems reasonable to adopt therapeutic strategies for these patients that are effective and easy to follow in the outpatient setting.

Cefditoren (CDN) is a third-generation cephalosporin for oral administration. CDN has a broad spectrum of activity and is particularly active against the bacterial pathogens involved in community respiratory tract infections. Besides that, the use of CDN has been associated with a marked decrease in circulating levels of IL-6 and other pro-inflammatory cytokines and mediators of epithelial damage. The aim of this study is to demonstrate that CDN improves clinical condition in patients with mild-moderate COVID-19 and symptoms of bacterial pneumonia.

DETAILED DESCRIPTION:
The global pandemic of novel coronavirus disease 2019 (COVID-19) began in Wuhan, China, in December 2019, and has since spread worldwide. The novel coronavirus is now referred to as severe and critical acute respiratory syndrome coronavirus-2 (SARS-CoV-2). The disease is mild in 85% of cases but the remaining 15% requires hospitalization and/or intensive care.

Recent publications show that a variable number of COVID-19 patients are co-infected with one or more pathogens. Most co-infections occurred within 1-4 days of onset of COVID-19 disease and in a retrospective study, secondary infection was observed in 50% of non-survivor patients.

In COVID-19 patients the elevated inflammatory cytokines and other inflammatory mediators present suggest that a cytokine storm, also known as cytokine release syndrome (CRS), may play a major role in the pathology of this disease. The elevated cytokine levels, specifically IL-6, may also be responsible for the lethal complications of COVID-19. Therefore, the interleukin-6 (IL-6) blockade has been proposed as one of the strategies to manage COVID-19-induced CRS.

A considerable number of COVID-19 patients arrive to the Emergency rooms with mild-moderate respiratory symptoms compatible with pneumonia of presumed bacterial origin not severe enough for requiring hospitalization. It therefore seems reasonable to adopt therapeutic strategies for these patients that are effective and easy to follow in the outpatient setting to avoid overloading the Health System.

Cefditoren (CDN) is a third-generation cephalosporin for oral administration. CDN has a broad spectrum of activity and is particularly active against the bacterial pathogens involved in community respiratory tract infections. The results of clinical trials with CDN on community-acquired pneumonia showed percentages of clinical and microbiological efficacy around 85%. On the other hand, the use of CDN has been associated with a marked decrease in circulating levels of IL-6 and other pro-inflammatory cytokines and mediators of epithelial damage such as Krebs von den Lungen-6 (KL-6).

Considering the above and the current estate of knowledge against SARS-CoV-2, we have considered of relevance to study the efficacy of CDN in a series of patients with mild-moderate COVID-19 and with symptoms compatible with pneumonia of presumed bacterial origin, seen at the Emergency room of a public hospital and followed on outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years
* Positive for SARS CoV-2
* Radiological and clinical signs of mild-moderate pneumonia
* Fever ≥37.7 ºC
* Sat O2> 94% and respiratory rate <24 on admission
* Able of taking oral medication
* HIV negative
* Written and signed consent

Exclusion Criteria:

* Concomitant treatments with drugs of demonstrated or potential action against SARS CoV-2 within the previous 24 hours.
* Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) > 5 times the upper limit
* corrected QT (QTc) interval prolongation> 450 msg,
* Moderate or severe renal impairment (creatinine<50ml/min)
* Severe hepatic impairment (Child-Pugh C)
* Pregnancy or childbearing
* Allergy to penicillin or any other beta-lactam
* Primary carnitine deficiency
* Malabsorption or swallowing problems
* Inability to understand and follow study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Evolution of patient status | 28 days
  Evolution of the status of the patient defined by the World Health Organization Ordinal Scale for Clinical Improvement for COVID-19. This is a 0-8 score where higher scores mean a better or worse outcome.
Assessment of Clinical improvement | 28 days
  Evaluation of clinical condition through a Clinical Improvement questionnaire.

SECONDARY OUTCOMES:
Additional visit to the Emergency room | 28 days
  New attendance to the hospital due to worsening
Need for hospitalization | 28 days
  Hospitalization due to worsening
Occurrence of adverse events | 28 days
  Adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Cristóbal Rodríguez Leal, Dr, Principal Investigator — HU Henares
Locations (1):
- HU Henares, Coslada, Madrid, Spain